CLINICAL TRIAL: NCT05102539
Title: Epidemiological Study of Non-invasive Fungal Sinusitis as Presented in Sohag University Hospital
Brief Title: Causes of Non-invasive Fungal Sinusitis as Presented in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Hafez Abd Elall, Principal Investigator at department of Otorhinolaryngology at sohag university, Sohag University
Other Study IDs: Soh-Med-21-09-08
Record Dates: First submitted 2021-10-04; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Sinus Infection
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
in this study, the investigators will collect data from patients with non-invasive fungal sinusitis to know what causes it

DETAILED DESCRIPTION:
In this study, the investigators will try to know the epidemiology of noninvasive fungal sinusitis, especially in recurrent cases This study will be carried out at sohag university hospital. Retrospective study Study period: 5 years (from August 2016 to August 2021. )

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute fungal sinusitis.
* Patients with chronic granulomatous sinusitis.
* Patients with sinus mycetomas.

Exclusion Criteria:

* Immunocompromised patients.
* invasive fungal sinusitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-invasive Fungal Sinusitis patients as Presented in Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
risk factors related to non-invasive fungal sinusitis | 5 years study period from august 2016 to august 2021
  retrospective study assessed by Statistical Package for Social Sciences

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes